CLINICAL TRIAL: NCT06422702
Title: A Prospective, Randomized, Single-blind Study on the Effects of Psychosomatic Symptom Interventions on Patients With Differentiated Thyroid Cancer During the Initial Treatment Period
Brief Title: The Effect of a Psychosomatic Symptom Intervention Program on the Primary Treatment of Differentiated Thyroid Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Shuhua Luo, researcher, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HMUDQ20231116204; 72004047 (Other Grant/Funding Number: National Natural Science Foundation of China); JFCX202303 (Other Grant/Funding Number: Fundamental Research Funds for the Provincial Universities，Heilongjiang,China); YJSCX2023-295HYD (Other Grant/Funding Number: Postgraduate Research & Practice Innovation Program of Harbin Medical University)
Record Dates: First submitted 2024-05-12; First posted 2024-05-21 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Pathologically Confirmed Differentiated Thyroid Carcinoma; All Patients Are in the Initial Treatment Phase; Normal Cognitive and Communicative Abilities, Capable of Reading and Understanding Questionnaires in Chinese; Ability to Use a Smartphone; Voluntary Participation in the Study and Signed Informed Consent
Keywords: Differentiated thyroid cancer; Anxiety; Depression; Thyroid stimulating hormone; Randomized block design
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): A 12-week psychosomatic symptom intervention was conducted
  Interventions: Other: Psychosomatic Symptoms Intervention
- control group (Other): Implementation of 12 weeks of continuous nursing (comfort attention)
  Interventions: Other: Extended supportive care

INTERVENTIONS:
Other: Psychosomatic Symptoms Intervention — Psychosomatic symptoms included intervention of negative psychological symptoms and intervention of physical discomfort symptoms.
  Arms: intervention group
Other: Extended supportive care — The control group implemented continuity of supportive care based on primary care
  Arms: control group

SUMMARY:
The psychosomatic symptoms of patients with differentiated thyroid cancer (DTC) during the initial treatment phase need to be improved. Stress coping training aims to reshape an individual's perception of stress and provide skill training, thereby influencing how they cope in stressful situations. Symptom management theory emphasizes improving health outcomes by helping individuals perceive and manage their symptoms.

Therefore, this clinical trial combines stress coping training and symptom management theory to construct and test an intervention program for psychosomatic symptoms in DTC patients. The main questions it aims to answer are:

* Does the psychosomatic symptom intervention alleviate participants' levels of anxiety and depression?
* Does the psychosomatic symptom intervention promote participants' achievement of TSH suppression therapy standards?
* Does the psychosomatic symptom intervention enhance participants' self-management efficacy?
* Does the psychosomatic symptom intervention improve participants' shoulder joint function?

Researchers will compare the psychosomatic symptom intervention with continuous psychological care (a form of comforting care) to determine if the intervention better promotes participants' psychosomatic health.

1. Before conducting this clinical trial, researchers conducted qualitative interviews with DTC patients and healthcare providers, followed by literature analysis and expert consultations to develop a psychosomatic symptom intervention program for DTC patients during the initial treatment phase.
2. A total of 84 DTC patients in the initial treatment phase were recruited and randomly grouped into two blocks. The intervention group received a 12-week psychosomatic symptom intervention in addition to routine care, while the control group received 12 weeks of continuous care. Data were collected before the intervention, at the end of the intervention, 3 months after the intervention, and 6 months after the intervention.

The psychosomatic symptom intervention mainly includes:

* Psychological module: symptom logs, meditation, positive psychology, and emotional management
* Physiological module: gargling exercises, "T" exercises, "米" exercises, and shoulder-neck exercises
* The psychosomatic module aims to intervene at three levels: individual, environmental, and health and disease. The individual level includes role management and self-awareness. The environmental level includes resource utilization, family support, peer support, and social support. The health and disease level includes disease management, individual counseling, and progressive muscle relaxation training.
* The intervention is divided into three stages: concept formation, skill acquisition and repetition, and application and completion. These stages are further divided into six sub-stages, each containing content from the psychological, physiological, and psychosomatic modules.

ELIGIBILITY:
Inclusion criteria:

1. Clinical diagnosis of differentiated thyroid cancer
2. Participants had to be in the initial treatment phase
3. Cognitive and communication skills are normal
4. Can use a smartphone
5. Voluntary participation in the study

Exclusion criteria:

1. History of neck or shoulder trauma
2. Coexisting serious heart, brain, or lung diseases
3. History of a major psychological disorder or mental illness
4. Patients taking hypnotics or psychotropic medications
5. have recently participated in a similar intervention or are receiving other psychotherapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2025-04-22 (Estimated)

PRIMARY OUTCOMES:
anxiety and depression | Before the beginning of the intervention (T0), at the end of the intervention (12 weeks of intervention, T1), and 3 and 6 months after the end of the intervention (T2 and T3).
  The Hospital Anxiety and Depression Scale (HADS) was used to assess the anxiety and depression levels of DTC patients. The scale was developed by Zigmond in 1983 and is primarily used to assess the anxiety and depression of the subjects over the past month. A total of 14 items were included, comprising an anxiety subscale and a depression subscale, each containing 7 items. According to the frequency of occurrence, the situation is divided into four levels, namely "1 to 4", scored from 0 to 3 points, and the two subscales range from 0 to 21 points. The lowest possible score is 0, while the highest is 42. Higher scores on the scale indicate more severe levels of anxiety and depression.

SECONDARY OUTCOMES:
TSH | Before the start of the intervention (T0), at the end of the intervention (up to 12 weeks of intervention, i.e., three months postoperatively, T1), and six months after the end of the intervention (i.e., nine months postoperatively, T2).
  This study is based on the recommended by 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer. First, in patients with a structural incomplete response to therapy, the serum TSH should be maintained below 0.1 mU/L. Secondly, in patients with a biochemical incomplete response to therapy, the serum TSH should be maintained between 0.1 and 0.5 mU/L. In patients with an excellent (clinically and biochemically free of disease) or indeterminate response to therapy, the serum TSH may be kept within the low reference range (0.5-2 mU/L). Finally, in patients who have not undergone remnant ablation, the serum TSH can be allowed to rise to the low reference range (0.5-2 mU/L).
Self-management efficacy | Before the beginning of the intervention (T0), at the end of the intervention (12 weeks of intervention, T1), and 3 and 6 months after the end of the intervention (T2 and T3).
  The Chinese version of Strategies Used by People to Promote Health (C-SUPPH) was used to evaluate the self-management efficacy of DTC patients. The scale was developed in 1996, and the Chinese version was revised by Huijuan Qian et al. There were 28 items in total, including 3 dimensions of positive attitude (items 7, 15 to 28), self-decision-making (items 10 to 12) and self-decompression (items 1 to 6, 8, 14). Each item was scored using the Likert 5 scale, with a score of 1 indicating no confidence and a score of 5 indicating very confident. The total score ranged from 28 to 140, ranging from 0 to 55 (low level), from 55 to 112 (medium level), and from >112 (high level), with higher scores indicating greater confidence in the individual to perform self-care.
Shoulder function | Before the beginning of the intervention (T0), at the end of the intervention (12 weeks of intervention, T1), and 3 and 6 months after the end of the intervention (T2 and T3).
  The Constant-Murley Shoulder Function Scale (CMS) was used to assess the shoulder joint activity of the two groups. The scale includes two dimensions: subjective evaluation and objective evaluation. Subjective evaluation included pain levels and activities of daily living. Objective evaluation included assessing shoulder range of motion and muscle strength. The lowest score is 0, the highest score is 100, higher scores indicate better shoulder function.

CONTACTS AND LOCATIONS:
Locations (1):
- Harbin Medical University, Harbin, Heilongjiang, China

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT06422702/Prot_SAP_ICF_000.pdf